CLINICAL TRIAL: NCT03658551
Title: Confocal Endoscopy to Diagnose the Intestinal Permeability in Patients With Compensated and Decompensated Liver Cirrhosis
Brief Title: Intestinal Permeability in Patients With Liver Cirrhosis Using Confocal Endoscopy
Acronym: CEDIP-LCI
Status: Terminated | Type: Observational
Why Stopped: Inability to apply technology (Loss of technology)
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Jörn M. Schattenberg, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: CEDIP_LCI_JGU
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Cirrhosis, Liver
Keywords: Portal hypertension; Intestinal permeability; Liver cirrhosis; bacterial translocation; confocal endoscopy
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Fluorescein Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue biopsy, serum, EDTA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Liver cirrhosis: Patients with liver cirrhosis are included in this arm. Liver cirrhosis is diagnosed by ultrasound, CT - scan oder by clinical signs.
  Interventions: Diagnostic Test: Fluorescein
- Control group: Patients with abdominal symptoms with the indication for endoscopy without liver cirrhosis and portal Hypertension.
  Interventions: Diagnostic Test: Fluorescein

INTERVENTIONS:
Diagnostic Test: Fluorescein — Measurement of intensity in the gastrointestinal mucosa after intravenous administration of fluorescein by confocal endoscopy
  Other Names: Intravenous application of fluorescein

SUMMARY:
The CEDIP LCI study is intended to show the difference in intestinal permeability between compensated and decompensated liver cirrhosis by confocal endoscopy.

DETAILED DESCRIPTION:
Liver cirrhosis often represents the end of many different liver diseases. A progress of liver cirrhosis with development of bleeding and infection complications represents a significant burden on the health system. It is therefore more important that the molecular basis leading to progress of liver cirrhosis is studied. In the last few years it has been demonstrated in various animal models as well as in human studies that the liver via the portal vein circuit is constantly under the influence of macronutrients, toxins, microbial products and microorganisms from the gastrointestinal tract. Patients with hepatic cirrhosis suffer from increased intestinal permeability so that bacterial components, endotoxins and pathogens enter the portal vein circuit via mesenteric lymph nodes. Bacterial translocations were found in patients with advanced liver cirrhosis and restricted organ function. This translocation causes a local as well as systemic inflammation with an increase in portal hypertension and further deterioration of the hepatic function, as well as a hyperdynamic circulatory situation which in many cases can lead to the death of the patient. These findings on the pathogenesis of portal hypertension and complications of cirrhosis of the liver have already led to the first therapeutic approaches where the occurrence of hepatic encephalopathy could be reduced by a purely intestinal reduction of the bacterial load by the antibiotic rifaxamine.

The intestinal barrier describes a functional and physical unit that ensures regulated intraluminal transport and protects against microorganisms and other pathogenic molecules. In addition to the intestinal epithelium with superposed mucus, intercellular proteins constitute an essential component. These paracellular proteins include tight junctions, anchoring junctions and GAP junctions, which are also responsible for controlled paracellular transport.

The cause of increased intestinal permeability in patients with liver cirrhosis are manifold. In addition to altered microbial colonization and slowed intestinal transit time, structural changes in the intestinal wall and altered expression of the tight junctions.

Due to the increasing insight into the molecular pathogenesis of intestinal permeability including portal hypertension, it is necessary to quantify these parameters more precisely in the clinical routine and to develop possible therapeutic interventions therefrom. An endoscopic procedure is provided by confocal endoscopy, with the aid of which portal hypertension and intestinal permeability can be diagnosed and estimated. With the help of this clinical study, this procedure is to be established.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* need of upper endoscopy
* signed consent
* abdominal symptoms with indication for endoscopy

Exclusion Criteria:

* pregnancy
* Lactation
* Hypersensitivity to fluorescein
* Limited coagulation situation (Quick <50%, PTT> 50 sec, thrombocyte count <50000 / μl or disturbed thrombocyte function) despite the substitution of coagulation factors / plasma products
* Limited or non-existent consent
* Restricted or inadequate ability to perform endoscopy and / or confocal imaging: restlessness of the patient, food residues, anatomical variants that make confocal imaging difficult (e.g., strictures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Amount of intestinal permeability | August 2020
  Intensity of fluorescein concentration in the gastrointestinal mucosa

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center of the Johannes Gutenber Univeristy, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Undecided